CLINICAL TRIAL: NCT07155564
Title: Energy Balance Within a Whole-Room Indirect Calorimeter and Its Relevance for Energy Expenditure Measures
Brief Title: Validation of Energy Expenditure Measures Study
Acronym: ValEE
Status: Recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: Helmholtz Center Munich (Unknown); University of Pisa (Other)
Responsible Party: Principal Investigator, Sascha Heinitz, Physician, University of Leipzig
Other Study IDs: 121-24/ek
Record Dates: First submitted 2025-01-20; First posted 2025-09-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-02

CONDITIONS: Obesity Prevention; Healthy
Keywords: Energy balance; Energy expenditure; Weight change; Energy intake; Indirect calorimetry
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy: Healthy subjects of both sexes meeting inclusion criteria.

SUMMARY:
The energy that the human body burns and the amount of food consumed determine a person's body weight. If food intake covers the amount of energy burned, body weight remains constant - a state known as energy balance. Achieving an energy balance is not easy in everyday life. This is reflected in the increasing number of people suffering from morbid obesity. To counteract this development, it is important to have a better understanding of how much food a person should eat.

In this study, the investigators will investigate the amount of food needed to meet a person's energy needs and bring them into energy balance.

Primary aims of the study are i) to technically and biologically validate two whole-room indirect calorimeters (WRICs) and ii) by using whole-room indirect calorimetry, to achieve a more accurate estimate of a person's emergy balance compared to common approximation formulas.

Secondary study aims:

1. To investigate whether the transfer of a person into energy balance using WRIC has an influence on energy expenditure measures compared to the transfer into energy balance using the usual approximation formula.
2. To investigate whether the transfer of a person into energy balance using WRIC has an influence on activity-dependent energy expenditure measures compared to the transfer into energy balance using the usual approximation formula.
3. To investigate whether differences in energy expenditure during energy balance during moderate and strenuous physical activity influence food intake.
4. To investigate whether energy intake in relation to energy expenditure during energy balance is related to weight development

DETAILED DESCRIPTION:
Technical Validation: Eight 24-hour methanol burns within each of the two WRICs will be conducted for technical validation.

Biological Validation and Energy Balance Component:

After providing informed consent and meeting inclusion/exclusion criteria, study participants will follow a weight-maintaining diet before their first 24-hour stay in a WRIC (Day 4). During this stay, energy expenditure will be measured under conditions of estimated energy balance. As a measure of energy expnediture relative to energy intake, energy balance will be estimated based on resting energy expenditure, an estimated physical activity level, and an approximation formula applied during the screening procedure.

A second 24-hour stay in the WRIC (Day 6), also under conditions of estimated energy balance, will serve for biological validation. After following the weight-maintaining diet for three additional days, a third 24-hour WRIC stay (Day 10) will assess the achievement of near-perfect energy balance. On the day following this stay (Day 11), participants will have access to a buffet and will be allowed to eat ad libitum.

Subsequently, a 3-day run-in period under weight-maintenance conditions will precede reassessment of 24-hour energy expenditure during increased physical activity in the WRIC (Days 15 and 17). Energy expenditure during energy balance will again be compared to ad libitum food intake at a buffet (Day 18).

Follow-up weight measurements will be conducted one year after study completion to evaluate the influence of achieving near-perfect energy balance-or deviations from it-on weight change. Additionally, fasting blood samples will be collected before and after each WRIC stay, as well as before and after ad libitum food intake, to measure hormones related to appetite control and satiety.

N = 34 subjects are required to detect a statistically significant difference in energy balance after measuring energy expenditure using a WRIC. However, interim analysis after n = 8 subjects will be conducted to adjust needed sample size to variability as detected using here implied methods of indirect calorimetry.

The statistical evaluation with regard to i) technical validation, ii) biological validation, and iii) testing the achievability of an energy balance and its effect on energy consumption are carried out using parametric and non-parametric tests. Data are given as mean value with standard deviation. The significance level is P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Abilty to provide informed consent
* Written declaration of consent
* Healthy study participants
* Able to perform moderate physical exercise using a bike ergometer
* Women: continuous contraception/fullicular phase of menstrual cycle

Exclusion Criteria:

* Weight change > 5 kg or 5% of body weight in the last 3 months
* Nicotine abuse, Alcohol/drug abuse
* Strenuous physical activity in everyday life > 1 h per day
* Body mass index < 18.5 kg/m² or ≥ 40 kg/m²
* Chronic diseases with an impact on energy expenditure
* Food allergy/intolerance, vegan diet
* Circumstances that speak against the application of wearable accelerometers (e.g. silicone contact allergy)
* Impaired fasting glucose, diabetes mellitus and prediabetes
* Pregnancy/breastfeeding
* Claustrophobia
* Refusal to communicate incidental findings

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Cisgender subjects
Study Population: Healthy, non-obese subjects of both sexes.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure | From enrollement to the end of 5th stay within the whole-room indirect calorimeter, study day 18.
  Repeated assessment of energy expenditure in the setting of a whole-room indirect calorimeter and relative to prior energy expenditure assessment using the ventilated hood method (canopy) and estimation formula.
Energy intake | From enrollement to the end of 5th stay within the whole-room indirect calorimeter, study day 18.
  Repeated assessment of energy intake in the setting of a whole-room indirect calorimeter and relative to prior energy expenditure assessment using the ventilated hood method (canopy) and estimation formula.
Coefficient of variation | Prior to enrollement of subjects (technical validation). From enrollement to the end of second stay within the whole-room indirect calorimeter, study day 7.
  Technical and biological validation via repeated assessment of methanol combustion as well as repeated stays within the whole-room indirect calorimeters. Measures: recovery, accuracy, macronutrient oxidation rates, respiratory exchange ratio, energy expenditure measures.

SECONDARY OUTCOMES:
Energy expenditure | From enrollement to the end of 5th stay within the whole-room indirect calorimeter, study day 11.
  Compared to common approximation formulas, achieving near perfect energy balance using a WRIC has an influence on energy expenditure measures (i.e. 24-hour energy expenditure, sleeping energy expenditure, diet-induced thermogenesis/awake-and-fed thermogenesis, physical exercise energy expenditure)
Physical exercise expenditure | From enrollement to the end of 5th stay within the whole-room indirect calorimeter, study day 18.
  Compared to common approximation formulas, achieving near perfect energy balance using a WRIC has an influence on energy expenditure measures in the setting of increased physical activity (i.e. 24-hour energy expenditure, sleeping energy expenditure, diet-induced thermogenesis/awake-and-fed thermogenesis, physical exercise energy expenditure)
Concentrations of hormones involved in energy intake | From enrollement to the end of 5th stay within the whole-room indirect calorimeter, study day 18.
  (Deviation from) near perfect energy balance relates to ad libitum energy intake and changes in hormones implied in appetite control/satiety. Outcome measures: ad libitum food intake during buffet, Leptin, Ghrelin, thyroid hormones, Cortisol, Insulin, IGF-1, Adiponectin, FGF21)
Body weight change | From enrollement to the end of 5th stay within the whole-room indirect calorimeter, study day 18. Body weight change follow-up one year after completion of the study.
  (Deviation from) near perfect energy balance relates to body weight change.

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Heinitz, MD, Principal Investigator — University of Leipzig
Locations (1):
- Department of Internal Medicine, Clinic for Endocrinology, Nephrology and Rheumatology, University of Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
The decision not to share IPD is based on considerations of participant privacy and data protection. Although all data are anonymized, the sensitive nature of the information collected in this study necessitates careful handling to minimize any risk of identification. Furthermore, the informed consent provided by participants does not explicitly include provisions for data sharing beyond the current study.
  To ensure compliance with ethical guidelines and data protection regulations, the study team has decided not to make IPD available publicly or to external researchers. However, summary data and study findings will be shared through peer-reviewed publications, ensuring transparency and the opportunity for scientific discourse.

REFERENCES:
- [Background] Stinson EJ, Rodzevik T, Krakoff J, Piaggi P, Chang DC. Energy expenditure measurements are reproducible in different whole-room indirect calorimeters in humans. Obesity (Silver Spring). 2022 Sep;30(9):1766-1777. doi: 10.1002/oby.23476. Epub 2022 Aug 3. PMID 35920141
- [Background] Piaggi P, Krakoff J, Bogardus C, Thearle MS. Lower "awake and fed thermogenesis" predicts future weight gain in subjects with abdominal adiposity. Diabetes. 2013 Dec;62(12):4043-51. doi: 10.2337/db13-0785. Epub 2013 Aug 23. PMID 23974925
- [Background] Weyer C, Snitker S, Rising R, Bogardus C, Ravussin E. Determinants of energy expenditure and fuel utilization in man: effects of body composition, age, sex, ethnicity and glucose tolerance in 916 subjects. Int J Obes Relat Metab Disord. 1999 Jul;23(7):715-22. doi: 10.1038/sj.ijo.0800910. PMID 10454105
- [Background] Hollstein T, Ando T, Basolo A, Krakoff J, Votruba SB, Piaggi P. Metabolic response to fasting predicts weight gain during low-protein overfeeding in lean men: further evidence for spendthrift and thrifty metabolic phenotypes. Am J Clin Nutr. 2019 Sep 1;110(3):593-604. doi: 10.1093/ajcn/nqz062. PMID 31172178
- [Background] Reinhardt M, Thearle MS, Ibrahim M, Hohenadel MG, Bogardus C, Krakoff J, Votruba SB. A Human Thrifty Phenotype Associated With Less Weight Loss During Caloric Restriction. Diabetes. 2015 Aug;64(8):2859-67. doi: 10.2337/db14-1881. Epub 2015 May 11. PMID 25964395
- [Background] Heinitz S, Hollstein T, Ando T, Walter M, Basolo A, Krakoff J, Votruba SB, Piaggi P. Early adaptive thermogenesis is a determinant of weight loss after six weeks of caloric restriction in overweight subjects. Metabolism. 2020 Sep;110:154303. doi: 10.1016/j.metabol.2020.154303. Epub 2020 Jun 27. PMID 32599082
- [Background] Ravussin E, Lillioja S, Anderson TE, Christin L, Bogardus C. Determinants of 24-hour energy expenditure in man. Methods and results using a respiratory chamber. J Clin Invest. 1986 Dec;78(6):1568-78. doi: 10.1172/JCI112749. PMID 3782471
- [Background] Venti CA, Votruba SB, Franks PW, Krakoff J, Salbe AD. Reproducibility of ad libitum energy intake with the use of a computerized vending machine system. Am J Clin Nutr. 2010 Feb;91(2):343-8. doi: 10.3945/ajcn.2009.28315. Epub 2009 Nov 18. PMID 19923376
- [Background] Weise CM, Hohenadel MG, Krakoff J, Votruba SB. Body composition and energy expenditure predict ad-libitum food and macronutrient intake in humans. Int J Obes (Lond). 2014 Feb;38(2):243-51. doi: 10.1038/ijo.2013.85. Epub 2013 May 23. PMID 23736368
- [Background] Basolo A, Votruba SB, Heinitz S, Krakoff J, Piaggi P. Deviations in energy sensing predict long-term weight change in overweight Native Americans. Metabolism. 2018 May;82:65-71. doi: 10.1016/j.metabol.2017.12.013. Epub 2018 Jan 3. PMID 29305947
- [Background] Hall KD, Heymsfield SB, Kemnitz JW, Klein S, Schoeller DA, Speakman JR. Energy balance and its components: implications for body weight regulation. Am J Clin Nutr. 2012 Apr;95(4):989-94. doi: 10.3945/ajcn.112.036350. No abstract available. PMID 22434603